CLINICAL TRIAL: NCT01949493
Title: Study of the Effectiveness of Mechanical Traction as a Non-Surgical Treatment for Carpal Tunnel Syndrome Compared to Care as Usual: a Randomized Controlled Trial
Brief Title: Non-surgical Treatment of Carpal Tunnel Syndrome by Means of Mechanical Traction
Acronym: MT-CTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tilburg University (Other)
Responsible Party: Principal Investigator, prof.dr. Victor J Pop, Prof. Dr. V.J.M. Pop, Tilburg University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL44692.008.13
Record Dates: First submitted 2013-09-19; First posted 2013-09-24 (Estimated); Last update posted 2016-12-09 (Estimated); Status verified 2016-12

CONDITIONS: Carpal Tunnel Syndrome
Keywords: carpal tunnel syndrome; traction; mechanical traction; Phystrac
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Care as usual (Other): The patient will receive the usual care provided by the neurologists at VieCuri Medical Center. This may include an expectant strategy, a wrist splint, corticosteroid injection or carpal tunnel release surgery.
  Interventions: Other: Care as usual
- Mechanical traction (Experimental): Twelve treatments with mechanical traction using the Phystrac traction apparatus.
  Interventions: Device: mechanical traction

INTERVENTIONS:
Device: mechanical traction — Twelve treatments with mechanical traction using the Phystrac traction apparatus. The Phystrac provides traction to the wrist using weights between 1 and 18 kg. The weights provide a pulling force in line with the forearm. After 8 seconds the weight is lifted, and there is a rest period of 4 seconds. This cycle will be repeated 10 times. Another two sets of 10 traction movements will be applied with the wrist positioned in 30 degrees supination and 30 degrees pronation. In total, 30 traction movements will be applied during each treatment.
  Other Names: Phystrac mechanical traction device (type GR 10)
  Arms: Mechanical traction
Other: Care as usual — Usual care provided by the neurologist (e.g. corticosteroid injection, wrist splint, carpal tunnel release surgery).
  Arms: Care as usual

SUMMARY:
The objective of this study is to evaluate the effectiveness of mechanical traction in patients with Carpal Tunnel Syndrome compared to care as usual.

DETAILED DESCRIPTION:
This randomized controlled trial will examine the effectiveness of mechanical traction compared to care as usual as a non-surgical treatment for Carpal Tunnel Syndrome (CTS).

Patients diagnosed with CTS are recruited from the outpatient neurology clinic of VieCuri Medical Center in Venlo, The Netherlands. They will be randomly assigned to the intervention or control group. Patients in the intervention group will receive 12 treatments with mechanical traction during six consecutive weeks. Patients in the control group will receive care as usual, which can include splinting, a corticosteroid injection, carpal tunnel release surgery or an expectant strategy. Outcomes will be assessed at baseline and at 3, 6, and 12 months after inclusion.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with CTS using electrodiagnostic testing
* being physically capable of visiting the outpatient clinic in Venlo twice per week
* being physically capable of sitting in upright position in a chair for 10-20 minutes, twice per week
* not intending to move outside the area within 3 months after inclusion

Exclusion Criteria:

* not understanding Dutch appropriately
* other known (rare) cause of neuropathy
* suffering from severe psychiatric disorders, such as personality disorder, schizophrenia or bipolar disorder

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2013-10; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in symptom severity and functional status on the Boston Carpal Tunnel Questionnaire (BCTQ) at 12 months | Baseline, 3 and 6 weeks (intervention group) and 3, 6 and 12 months.
  Functional status and symptom severity will be measured using a self-reported scale: the BCTQ. The BCTQ is a disease-specific questionnaire and consists of two different scales: the Symptom Severity Scale (SSS) and the Functional Status Scale (FSS). The SSS consists of 11 questions about symptom severity. The FSS consists of 8 daily activities which are rated based on degree of difficulty. The SSS and the FSS are rated on a five-point scale, where a higher score represents a greater impairment.

SECONDARY OUTCOMES:
Change from baseline in quality of life on abbreviated version of the World Health Organisation Quality of Life (WHOQOL-BREF) | Baseline, 6 weeks (intervention group) and 3, 6 and 12 months.
  Self-reported quality of life will be measured using the WHOQOL-BREF in Dutch. It consists of 26 items which can be scored on a five-point scale. Better quality of life is represented by a higher score.
Change from baseline in absenteeism from work | Baseline, 3 and 6 weeks (intervention group) and 3, 6 and 12 months.
  A non-standardized questionnaire is used to collect the number of days off work of each patient. Patients are also asked if they are currently on sick leave or have been because of their CTS complaints.
Change from baseline in health care related resource utilization | Baseline, 3 and 6 weeks (intervention group) and 3, 6 and 12 months.
  A non-standardized questionnaire is used to assess if patients have visited a professional caregiver (general practitioner, physiotherapist, psychologist, etc.) in the past 12 months, if they spent time in the hospital or use medication.

OTHER OUTCOMES:
Change from baseline in depression and anxiety on the 4-item Patient Health Questionnaire (PHQ-4) | Baseline, 6 weeks (intervention groups and 3, 6, and 12 months.
  Self-reported depression and anxiety is measured using the PHQ-4. The questionnaire consists of 2 items on depression and 2 on anxiety answered on a 4-point scale, where a higher score represents a higher level of anxiety and depression.

CONTACTS AND LOCATIONS:
Overall Officials: Victor Pop, Prof. Dr., Principal Investigator — Tilburg University
Locations (1):
- Viecuri Medisch Centrum, Venlo, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Meems M, Boekhorst MGBM, Pop VJM. Long-Term Follow-Up Results of Mechanical Wrist Traction as Non-Invasive Treatment for Carpal Tunnel Syndrome. Front Neurol. 2021 Sep 6;12:668549. doi: 10.3389/fneur.2021.668549. eCollection 2021. PMID 34552548